CLINICAL TRIAL: NCT01232244
Title: Oxyntomodulin, Mechanisms of Action in Relation to Appetite, Food Intake, Gastric Emptying and Energy Expenditure.
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Jonatan I Bagger, MD, University Hospital, Gentofte, Copenhagen
Other Study IDs: OXMDissek
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Incretin Action; Obesity
Keywords: Incretin hormones; Glucagon; Satiety; Hunger; Energy expenditure
MeSH Terms: conditions — Obesity | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy young males
  Interventions: Other: GLP-1 infusion; Other: Glucagon infusion; Other: Oxyntomodulin infusion; Other: GLP-1 and glucagon infusion; Other: Placebo

INTERVENTIONS:
Other: GLP-1 infusion — 1 pmol/kg/min
Other: Glucagon infusion — 3ng/kg/min
Other: Oxyntomodulin infusion — 3 pmol/kg/min
Other: GLP-1 and glucagon infusion — 1 pmol/kg/min 3 ng/kg/min
Other: Placebo — NaCl 9 g/L infusion

SUMMARY:
Tiny molecules (hormones) are released from the bowels and other organs to the bloodstream in response to meals in order to orchestrate the metabolism. Oxyntomodulin, GLP-1 and glucagon are all known to regulate parameters such as appetite, food intake and induce weight loss.

Therefore we want to investigate mechanistic relations between the three hormones.

ELIGIBILITY:
Inclusion Criteria:

* Normal fasting plasma glucose
* Normal glucose tolerance
* Normal haemoglobin levels
* Informed content

Exclusion Criteria:

* Diabetes
* Pre diabetes (impaired glucose tolerance or impaired fasting glucose)
* 1st degree relatives with diabetes
* Obesity (BMI > 30)
* Inflammatory bowels disease
* Bowels surgery
* Nephropathy
* Liver disease
* Medication which cannot be on hold for 24h

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy young males
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Gastric emptying | 4 h
  Assessed by the acetaminophen - method
Satiety | 4 h
  Assessed by VAS
Hunger | 4 h
  Assessed by an ad'libitum meal
basal energy expenditure | 2 x 30min
  Assessed by indirect calorimetry

SECONDARY OUTCOMES:
GLP-1 | 4 h
Oxyntomodulin | 4 h
Glucagon | 4 h
GIP | 4 h

CONTACTS AND LOCATIONS:
Overall Officials: Jonatan I Bagger, MD, Principal Investigator — Gentofte University Hospital, University of Copenhagen
Locations (1):
- Gentofte University Hospital, Hellerup, Denmark

REFERENCES:
- [Derived] Bagger JI, Holst JJ, Hartmann B, Andersen B, Knop FK, Vilsboll T. Effect of Oxyntomodulin, Glucagon, GLP-1, and Combined Glucagon +GLP-1 Infusion on Food Intake, Appetite, and Resting Energy Expenditure. J Clin Endocrinol Metab. 2015 Dec;100(12):4541-52. doi: 10.1210/jc.2015-2335. Epub 2015 Oct 7. PMID 26445112